CLINICAL TRIAL: NCT02922972
Title: Efficay of Autologous Platelet Rich Plasma Obtained With RgenKit-BCT in the Prevention and the Treatment of Keloid Scars
Brief Title: Treatment of Keloid Scar by Autologous Platelet Rich Plasma Obtained With RgenKit-BCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regen Lab SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-A00163-44
Record Dates: First submitted 2016-09-30; First posted 2016-10-04 (Estimated); Last update posted 2019-11-15 (Actual); Status verified 2019-11

CONDITIONS: Keloid
Keywords: Keloid scar; Wound healing; Platelet-Rich Plasma; RegenLab
MeSH Terms: conditions — Keloid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Platelet Rich Plasma (Experimental): Interventions: Four injections of PRP: The first injection of A-PRP after complete resection of the keloid scar,Three additional injections were administered with a one-month interval.
  Interventions: Device: Autologous Platelet Rich Plasma obtained with RegenKit®-BCT

INTERVENTIONS:
Device: Autologous Platelet Rich Plasma obtained with RegenKit®-BCT — After complete resection of the keloid scar, the first injection was administered before closure into the lesion resection bed and edges. Three additional injections were administered with a one-month interval.
  Other Names: RegenKit®-BCT

SUMMARY:
The aim of this prospective study is to assess the efficacy of autologous Platelet Rich Plasma prepared with RegenKit-BCT in the prevention and the treatment of keloid scars refractory to conventional treatments. Fifteen patients were included and received three PRP injection sessions with a one-month interval. The outcomes were assessed at baseline (before treatment), 3, 6, 12 and 24 months after the last injection session. Safety was assessed by reported adverse event analysis.

DETAILED DESCRIPTION:
To evaluate the efficacy and the safety of platelet rich plasma in the treatment of keloid scars. This prospective, comparative study (before-after treatment) included 15 patients with keloid scars refractory to conventional treatment (corticoids, surgery, cryotherapy). The primary outcome was the percentage of patients achieving a complete remission of their keloid scar 2 years after the end of treatment. Secondary outcomes were the Vancouver scar scale and pruritus severity scored at 3, 6, 12 and 24 months post treatment vs baseline.

ELIGIBILITY:
Inclusion Criteria:

* Patients with keloid scars refractory to conventional treatments. The indication of PRP injection was based on the absence of response to corticosteroids alone or in combination with surgery after 4 sessions of infiltration and/or absence of response to other therapies.

Exclusion Criteria:

* Patients younger than 18 years
* Pregnancy or breastfeeding
* Patients suffering from anemia
* patients with active skin disorder infection including active hepatitis or human infection virus infection
* Auto-immune disease such as Hashimoto, rheumatoid arthritis.
* Malignancy with or without metastatic disease
* Chemotherapy
* Anticoagulant therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Percentage of patients achieving a complete remission of their keloid scar 2 years after the end of treatment. | 24 months
  The efficacy of autologous platelet concentrate obtained with RegenKit®-BCT was assessed based on the percentage of patients achieving a complete remission of their keloid scar 2 years after the end of treatment.

SECONDARY OUTCOMES:
Evaluation of the scar using Vancouver scale. | 24 months
  The efficacy of the treatment was also assessed and determined using the Vancouver scar scale.
prirutis severity | 24 months
  The efficacy of the treatment was also assessed on the Pruritus severity
Pain assessment | 3 months
  pain assessment during injections were also scored using the VAS.
patient satisfaction | 24 months
  Patient satisfaction at the end of follow-up was assessed using a 0-10 VAS
Adverse events | 24 months
  Adverse events were reported.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hersant B, SidAhmed-Mezi M, Picard F, Hermeziu O, Rodriguez AM, Ezzedine K, Meningaud JP. Efficacy of Autologous Platelet Concentrates as Adjuvant Therapy to Surgical Excision in the Treatment of Keloid Scars Refractory to Conventional Treatments: A Pilot Prospective Study. Ann Plast Surg. 2018 Aug;81(2):170-175. doi: 10.1097/SAP.0000000000001448. PMID 29762444